CLINICAL TRIAL: NCT01049685
Title: Lopinavir/Ritonavir or Efavirenz as First-line Antiretroviral Therapy in Brazil: a "Real Life" Study
Brief Title: Lopinavir/Ritonavir or Efavirenz as First-line Antiretroviral Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Alexandre Naime Barbosa, SAE e Hospital Dia Domingos Alves Meira - Faculdade de Medicina de Botucatu - Unesp
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: upeclin/HC/FMB-Unesp-38
Record Dates: First submitted 2010-01-11; First posted 2010-01-14 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-01

CONDITIONS: HIV Infections
Keywords: HIV; Antiretroviral Therapy, Highly Active; Efavirenz; Lopinavir; Comparative Effectiveness Research; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — efavirenz; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Efavirenz Group (Active Comparator): Naïve-treatment HIV patients, who started therapy with Efavirenz
  Interventions: Drug: First-line Antiretroviral Therapy
- Lopinavir/r Group (Active Comparator): Naïve-treatment HIV patients, who started therapy with Lopinavir/ritonavir
  Interventions: Drug: First-line Antiretroviral Therapy

INTERVENTIONS:
Drug: First-line Antiretroviral Therapy — * Lopinavir/ritonavir: 02 capsules 12/12h, plus NRTI background
  * Efavirenz: 01 capsules day, plus NRTI background
  Other Names: Sustiva; Kaletra

SUMMARY:
Retrospective longitudinal cohort study with 36 HIV naïve-treatment patients, who started therapy with lopinavir/ritonavir or efavirenz (LPV/r or EFZ), follow-up of 36 months. Primary endpoint: virological success (HIV RNA <50 copies/mL) in the first six months and at the end of the study.

DETAILED DESCRIPTION:
Background: Either LPV/r or EFZ plus a two nucleoside reverse-transcriptase inhibitors (NRTIs) are recommended by the current guidelines all around the world as the main background drugs for initial therapy of human immunodeficiency virus type 1 (HIV-1) infection. This indication is based in results of clinical trials, but patients who participate in these studies usually are greatly motivated to continue their prescribed regimen, and can be different from the "real life". Therefore, clinical practice often cannot reproduce published results.

Methods: A retrospective longitudinal cohort study was performed with 36 naïve-treatment patients, who started therapy with LPV/r or EFZ, with follow-up of 36 months. The primary endpoint was virological success (HIV RNA <50 copies/mL) in the first six months and at the end of the study. Effectiveness was examined comparing time to virological failure and CD4 recovery.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected naive-treatment patients

Exclusion Criteria:

* use of Anti-Retroviral Agents in the past

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-08; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Maintenance HIV RNA <50 copies/mL at the end oh 36 months | 36 months

SECONDARY OUTCOMES:
Achieve HIV RNA <50 copies/mL at the first 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre N Barbosa, MD, MSc, Principal Investigator — Botucatu School of Medicine
Locations (1):
- SAE e Hospital Dia Domingos Alves Meira, Botucatu, São Paulo, Brazil